CLINICAL TRIAL: NCT02524964
Title: Effects of Sodium Tanshinone IIA Sulfonate on Left Ventricular Remodeling in Patients With ST-segment Elevation Myocardial Infarction Following Percutaneous Coronary Intervention
Brief Title: Sodium Tanshinone IIA Sulfonate in Left Ventricular Remodeling Secondary to Acute Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, shuai Mao, Department of Critical Care Medicine, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2014-011-01
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Left Ventricular Remodeling; Acute Myocardial Infarction
Keywords: left ventricular remodeling; cardiac magnetic resonance imaging; acute myocardial infarction
MeSH Terms: conditions — Ventricular Remodeling | interventions — tanshinone II A sodium sulfonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium tanshinone IIA sulfonate (Experimental): sodium tanshinone IIA sulfonate (80 mg q.d. for 7 days)
  Interventions: Drug: sodium tanshinone IIA sulfonate
- control (Sham Comparator): same volume/day of normal saline.
  Interventions: Other: control

INTERVENTIONS:
Drug: sodium tanshinone IIA sulfonate — eligible participants were randomized to receive sodium tanshinone IIA sulfonate injection (drip 80 mg/day for 7 days immediately after PCI)
  Other Names: sodium tanshinone IIA sulfonate injection
  Arms: sodium tanshinone IIA sulfonate
Other: control — equivalent volume of sodium chloride solution
  Other Names: sodium chloride solution
  Arms: control

SUMMARY:
Approximately 60 patients with ST-segment elevation myocardial infarction successfully treated with primary percutaneous coronary intervention will be enrolled and randomized to receive the sodium tanshinone IIA sulfonate in addition to standard therapy or the same volume/day of normal saline.

The primary endpoint is the variation in LV end-diastolic volume index (LVEDVi) assessed with cardiac magnetic resonance imaging (MRI) at baseline and 6 months.

DETAILED DESCRIPTION:
The primary endpoint is to determine whether sodium tanshinone IIA sulfonate could prevent LV remodeling among patients with completely reperfused AMI after PCI, detected by 6 month change in LVEDVi measured using cardiac MRI when compared to placebo.

Secondary endpoints will include cardiac MRI measures of variations in microvascular obstruction, defect size, ventricular wall motion score, wall thickening, global LV ejection fraction, ventricular volumes (LV end-systolic/ diastolic volume) and myocardial perfusion during the same interval.

Furthermore, the investigators will determine the variation (change from baseline) of biomarkers indicating myocardial fibrosis (PICP, PIIINP, ICTP and MMPs) and NT-ProBNP at 1 and 6 months after AMI.

Additional efficacy endpoints will include 6-minute walk test, New York Heart Association functional classification, Seattle Angina Questionnaire score and incidence of cardiovascular events (defined as cardiogenic death, stroke, recurrent myocardial infarction, readmission on account of deterioration of congestive heart failure or unstable angina, target vessel revascularization) at the 6-month follow-up will also be analyzed to evaluate the efficacy of sodium tanshinone IIA sulfonate treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18 years or over and under 80 years;
* 2. First-time myocardial infarction on admission;
* 3. Presence of STEMI who has successfully coronary recanalization by PCI within 12 h after the symptom onset;
* 4. Willingness to provide informed consent prior to enrollment;
* 5. Patient is able to comply with all follow-up evaluation

Exclusion Criteria:

* 1. Contraindications to performance of CMRI [pacemakers, implantable cardioverter/defibrillator devices, cardiac resynchronization therapy (CRT), claustrophobia, metal implants (joint prosthesis, et al), history of penetrative eye lesion];
* 2. Previous myocardial infarction, arrhythmia (including atrial fibrillation or bundle brunch block), significant valvular disease, and hypertrophic cardiomyopathy;
* 3. Severe heart failure (NYHA cardiac function class IV or left ventricular ejection fraction≤30%) or cardiogenic shock;
* 4. Serious impairment of renal function (glomerular filtration rate ≤50 mL/min per 1.73 m2);
* 5. Hypohepatia (elevated of alanine aminotransferase and aspartate aminotransferase serum levels);
* 6. Severe coagulopathy prior to randomization;
* 7. Malignant tumors or other life-threatening diseases with limited life expectancy <1 year;
* 8. Significant neuropsychopathic condition precluding written informed consent;
* 9. Pregnant and lactating women;
* 10. Known radiographic contrast or sodium tanshinone IIA sulfonate allergy;
* 11. Be on therapy with immunosuppressants;
* 12. Currently participated in any other investigational therapeutic or device trial;
* 13. Clinical follow-up over the next half years not possible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
left ventricular end-diastolic volume index | 6 months
  The primary endpoint is to determine whether sodium tanshinone IIA sulfonate could prevent LV remodeling among patients with completely reperfused AMI after PCI, detected by 6 month change in left ventricular end-diastolic volume index (mL/m^2) measured using cardiac magnetic resonance imaging .

SECONDARY OUTCOMES:
cardiac magnetic resonance imaging measures of LV remolding | 6 months
  cardiac magnetic resonance imaging measures of variations in left ventricular end-systolic/ diastolic volume (mL) during the same interval.
cardiac magnetic resonance imaging measures of microvascular obstruction | 6 months
  cardiac magnetic resonance imaging measures of the frequency of delayed or absent wash-in of contrast agent into the infarct zone.
variation (change from baseline) of biomarkers indicating myocardial fibrosis | 6 months
  type 1 collagen telopeptide (ng/mL), aminoterminal propeptide of type I procollagen (ng/mL), aminoterminal propeptide of type III procollagen (ng/mL), matrix metalloproteinase2 (ng/mL), matrix metalloproteinase9 (ng/mL) at 1 and 6 months after AMI.
major adverse cardiac event | 1 and 6 months
  frequency of the reported cardiovascular events (defined as cardiogenic death, stroke, recurrent myocardial infarction, readmission on account of deterioration of congestive heart failure or unstable angina, target vessel revascularization)
6-minute walk test | 6 months
  A 6-minute walk test measures the distance patients can quickly walk in 6 minutes. (in meters)
New York Heart Association functional classification | 6 months
  I Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc.
  II Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Seattle Angina Questionnaire score | 6 months
  The Seattle Angina Questionnaire is a valid and reliable instrument that measures five clinically important dimensions of health in patients with coronary artery disease (physical limitation, anginal stability, anginal frequency, treatment satisfaction, and disease perception). (in Units on a Scale).

CONTACTS AND LOCATIONS:
Overall Officials: minzhouzhang zhang, M.D., Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Yang F, Wu Y, Lu J, Gao X, Zhu X, Yang J, Liu S, Xiao G, Pan X. Identification of tanshinone I as cap-dependent endonuclease inhibitor with broad-spectrum antiviral effect. J Virol. 2023 Oct 31;97(10):e0079623. doi: 10.1128/jvi.00796-23. Epub 2023 Sep 21. PMID 37732786
- [Derived] Mao S, Li X, Wang L, Yang PC, Zhang M. Rationale and Design of Sodium Tanshinone IIA Sulfonate in Left Ventricular Remodeling Secondary to Acute Myocardial Infarction (STAMP-REMODELING) Trial: A Randomized Controlled Study. Cardiovasc Drugs Ther. 2015 Dec;29(6):535-542. doi: 10.1007/s10557-015-6625-2. PMID 26482376